CLINICAL TRIAL: NCT03939182
Title: Phase I Study of Abexinostat and Ibrutinib in Diffuse Large B-cell Lymphoma and Mantle Cell Lymphoma
Brief Title: Abexinostat and Ibrutinib in Diffuse Large B-cell Lymphoma and Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Xynomic Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-080
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Large B-cell Lymphoma; Mantle Cell Lymphoma
Keywords: Abexinostat; Ibrutinib; 19-080
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — abexinostat; ibrutinib

STUDY DESIGN:
Intervention Model Description: This is a phase I with dose expansion, open label single institution trial. The first stage is a standard 3+3 dose escalation trial. In the second stage, the dose expansion cohort will accrue patients at the MTD abexinostat and ibrutinib previously determined.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abexinostat and Ibrutinib (Experimental): The investigational agents to be used in this study are ibrutinib and abexinostat. Ibrutinib will be administered once daily on a 28-day cycle. Abexinostat will be administered orally twice daily (approximately 4-6 hours apart) for 7 days a week given every other week on a 28-day cycle.
  Interventions: Drug: Abexinostat; Drug: Ibrutinib

INTERVENTIONS:
Drug: Abexinostat — Two doses of the abexinostat will be tested: 30 mg/m2 and 45 mg/m2 orally twice daily, 7 days/week given every other week during a 28-day cycle.
Drug: Ibrutinib — Ibrutinib will be given at the FDA-approved dose for mantle cell lymphoma (MCL) of 560 mg orally daily for 28 day cycle.

SUMMARY:
The purpose of this study is to test the safety of abexinostat at different doses to find out if it can work with ibrutinib to stop the cancer from growing.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age at the time of signing Informed Consent
* Patient is able and willing to adhere to the study visit schedule and other protocol requirements
* Patient has histologically confirmed diagnosis of R/R mantle cell lymphoma or diffuse large B cell lymphoma

  * Diffuse large B cell lymphoma patients must have received at least 1 prior regimen and received, declined, or is ineligible for autologous or allogeneic stem cell transplant.
  * Diffuse large B cell lymphoma patients must have non-germinal center subtype disease applying the Hans classification algorithm using immunohistochemistry markers CD10, BCL6, and MUM1 (8).
  * Mantle cell lymphoma patients must have received at least 1 line of therapy
  * Allogeneic stem cell transplant recipients be greater than 6 months post transplant, not on immunosuppression for prevention of graft versus host disease for >3 months and without active graft versus host disease
  * Autologous stem cell transplant recipients must have adequate bone marrow recovery and are transfusion independent
  * Patients with transformed DLBCL from an antecedent or simultaneous indolent B-cell Non-Hodgkin lymphoma are permitted.
* Patient has at least one measurable lesion (≥ 1.5 cm) according to RECIL
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patient has adequate bone marrow and organ function by:
* Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L independent of growth factor support
* Platelets ≥100 x 10^9/L independent of transfusion

  °For patients with documented bone marrow involvement of underlying MCL or DLBCL at time of study enrollment, platelets must be ≥75 x 10^9/L independent of transfusion
* Hemoglobin (Hgb) ≥ 9.0 g/dL

  °For patients with documented bone marrow involvement of underlying MCL or DLBCL at time of study enrollment, Hgb must be ≥ 8.0 g/dL
* International Normalized Ratio (INR) ≤ 1.5
* Creatinine clearance > 25 mL/min as determined by the Cockcroft-Gault equation or a 24-hour urine collection
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ ULN (or ≤3 x ULN if liver involved with disease Total serum bilirubin ≤ 1.5 ULN unless bilirubin rise is due to Gilbert"s syndrome or of non-hepatic origin
* Normal serum potassium level with or without supplementation.
* Left Ventricular Ejection Fraction (LVEF) ≥ 50%
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trial. For females, these restrictions apply for 30 days month after the last dose of study drug. For males, these restrictions apply for 120 days after the last dose of study drug. Refer to section 9.7 "Reproductive toxicity" for additional details
* Women of childbearing potential must have a negative urine pregnancy test at Screening and within 7 days of treatment initiation
* Men must agree to not donate sperm during and 12 months after the study. Women should not donate ova/ooctyes for the purposes of
* Patient is able to swallow and retain oral medications

Exclusion Criteria:

* Patients previously treated with ibrutinib or HDAC inhibitor
* Patient has a history of non-compliance to medical regimen or inability to grant consent
* Patient is concurrently using other approved or investigational antineoplastic agent
* Patient has not recovered to Grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
* Patient has had major surgery or a wound that has not fully healed within 4 weeks of starting study drugs.
* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study
* Patient has evidence of active graft versus host disease (GVHD)
* Patient has active central nervous system (CNS) disease or meningeal involvement.
* Patient has history of stroke or intracranial hemorrhage ≤ 6 months from starting study drugs.
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patient has clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification, Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO), unstable angina pectoris, symptomatic pericarditis, QTcF > 480 msec on the screening ECG (using the QTcF formula), or history of congenital long QT syndrome.
* Patient has a concurrent active malignancy.
* Malignancies treated with a curative intent with an expected life expectancy ≥ 5 years or a non-competing life expectancy risk are eligible (i.e. adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer, early stage breast cancer, treated prostate cancer or any other cancer from which the patient has been disease free for ≥ 3 years).
* Patient with known history of human immunodeficiency virus (HIV), or any uncontrolled active systemic infection.
* Patients with acute viral hepatitis or a history of chronic or active HBV or HCV infection.

  * Hepatisis B surface antigen and core antibody testing are required at screening. If Hepatisis B surface antigen is positive then HBV PCR is required and if positive, then patient will be excluded.
  * Hepatisis C antibody testing is required at screening. If positive, Hepatisis C PCR is required and if positive, pHepatisis C PCR is required and if positive, then patient will be excluded.
* Patient has hepatic failure (Child-Pugh Class C)
* Patient is currently receiving increasing or chronic treatment (> 10 days) with corticosteroids or another immunosuppressive agent. Patients requiring chronic therapy with steroids may take no more than 10mg daily of prednisone or equivalent.
* Patient requires chronic treatment with a strong cytochrome P450 (CYP) 3A4 inhibitors, and inducers, or drugs known to induce Torsades de Pointes and the treatment cannot be discontinued or switched to a different medication prior to starting study drug (Appendix 1 and 3).
* Patients with known bleeding diathesis (e.g. von Willebrand "s disease) or hemophilia
* Patient is currently receiving warfarin or other Vitamin K antagonist. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed. Refer to Section 9.5 for Concomitant medication
* Vaccinated with live, attenuated vaccines within 4 weeks of randomization
* Patients with any life-threatening illness, medical condition or organ system dysfunction that in the opinion of the investigator could compromise the subject"s safety, interfere with absorption of metabolism of study drugs or put the study outcomes at undue risk.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
the MTD of abexinostat when combined with ibrutinib | 1 year
  a standard 3+3 dose escalation scheme will be used. For any given dose an initial cohort of 3 patients will be treated at that dose. The dose level will be escalated if none of the 3 patients exhibits any DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Salles, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm